CLINICAL TRIAL: NCT03418246
Title: Gingival Health Around Cervical Carious Lesions Restored With Calcium Silicate Based Cement (Biodentine) Compared With Glass-ionomer Cement: A Randomized Clinical Trial
Brief Title: Cervical Carious Lesions Restored With Calcium Silicate Based Cement (Biodentine) Compared With Glass-ionomer Cement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Rola Abdelraheem Alhabashneh, Prof, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JordanUST5
Record Dates: First submitted 2018-01-06; First posted 2018-02-01 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Gingivitis
Keywords: gingiva; plaque; pocket depth
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: One group will be treated with a tooth colored filling that will be placed near the gum line (Glass Ionomer). The second group will be treated with Biodentine that will be placed near the gum line.
Who Masked: Participant, Investigator
Masking Description: Investigator and participants are blinded to restoration used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GIC filling (Sham Comparator): Intervention/treatment One group will be treated with a tooth colored filling that will be placed near the gum line (Glass Ionomer).
  Placebo Comparator: GIC
  Participants will have a restoration placed with GIC in the lesion near the gum line. Device: GIC Application of a tooth colored filling in the cavitated dental lesion. Other Name: Resin modified glass ionomer
  Interventions: Device: GIC
- Biodentine filling (Experimental): Intervention/treatment The second group will be treated with Biodentine that will be placed near the gum line.Experimental: Biodentine
  Participants will have a restoration placed with Biodentine in the lesion near the gum line. Device: Biodentine Application of a white colored filling in dental lesion.
  Interventions: Device: Biodentine

INTERVENTIONS:
Device: GIC — tooth colored filling
  Arms: GIC filling
Device: Biodentine — White filling -Biodentine
  Other Names: Calcium Cilicate
  Arms: Biodentine filling

SUMMARY:
This study will test if applying calcium silicate cements (Biodentine) to restore cervical carious lesions might adversely affect the gingival health in comparison with conventionally used tooth colored material (GIC)

DETAILED DESCRIPTION:
The study will compare two different dental materials on dental lesions near the gum line. . The study will determine if one material is more effective in gingival health, after the placement of the two different dental materials.The oral hygiene and the gingival health of the restored teeth will be evaluated clinically at 1, 3 and 6-month intervals.

ELIGIBILITY:
Inclusion Criteria:

1. good general health;
2. good oral hygiene; and
3. age range 18-60 years old.

Patients with the following criteria were excluded:

1. current smokers;
2. pregnant females;
3. or patient with periodontal diseases; and
4. those who had a history of poorly controlled diabetes, liver disease, malignancy, radiotherapy.

Exclusion Criteria:

1. Pregnant women
2. Patients taking benzodiazepines, narcotics and multiple antidepressants for pain management not associated with the oral cavity
3. Patients requiring treatment for more than 5 decayed sites, periodontal disease and root canal therapy
4. Complicated medical history (>4 concurrent treatment for systemic diseases)
5. Lesion >1mm below the gum line

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-01-03 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-12-28 (Actual)

PRIMARY OUTCOMES:
Changes in Gingival index around Cervical Carious Lesions Restored with Calcium Silicate Based Cement (Biodentine™) Compared with Glass-Ionomer Cement; | 6 months
  Gingival health will be measured using the Loe -Silness gingival scoring Index (1963) which scores gingivitis on a numerical scale according to the following criteria:
  * 0 = Absence of inflammation.
  * 1 = Mild inflammation, slight change in color, slight edema, no bleeding on probing.
  * 2 = Moderate inflammation, moderate glazing, redness, bleeding on probing.
  * 3- Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous
    * Gingival index will be evaluated at four sites (mesial, distal, buccal, and lingual) on each tooth
Changes in Plaque accumulation around Cervical Carious Lesions Restored with Calcium | 6 months
  detect plaque level around restorations Plaque index (PI) (Silness and Löe, 1964). Plaque levels was measured using the Plaque Index Silness and Loe in 1964
  Score Criteria
  0 No plaque
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth, which cannot be seen with the naked eye. But only by Using disclosing solution or by using probe.
  2. Moderate accumulation of deposits within the gingival pocket, on the gingival margin and/ or adjacent tooth surface, which can be seen with the naked eye.
  3. Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin. Plaque index will be evaluated at four sites (mesial, distal, buccal, and lingual) on each tooth

SECONDARY OUTCOMES:
Changes in Pocket Depth around Cervical Carious Lesions Restored with Calcium | 6 months
  Probing depths (PD) will be measured at six sites (mesial, distal, and middle sites of the buccal and lingual sides) on each tooth using a Williams periodontal probe. PD will be measured from gingival margin to the base of the pocket.

CONTACTS AND LOCATIONS:
Overall Officials: Rola Al Habashneh, ABP, Study Director — JUST

IPD SHARING:
Plan to Share IPD: No